CLINICAL TRIAL: NCT00239213
Title: A Randomized Clinical Study of Catechin Gargling Effects on the Prevention of Influenza Infection
Brief Title: Catechin Gargling for Influenza Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Shizuoka (Other)
Collaborators: Shizuoka General Hospital (Unknown); Seirei Hamamatsu General Hospital (Other); White Cross Nursing Home (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CT2005002
Record Dates: First submitted 2005-10-13; First posted 2005-10-14 (Estimated); Last update posted 2006-10-31 (Estimated); Status verified 2006-10

CONDITIONS: Influenza Infection
Keywords: catechins; gargling; healthy volunteers

INTERVENTIONS:
Drug: catechin extracts (health food)

SUMMARY:
The purpose of this study is to clarify the preventive effects of catechin gargling on the influenza infection.

DETAILED DESCRIPTION:
In-vitro experimental studies have revealed that tea catechin extracts induce preventive effects on influenza infection. However, few studies have been conducted on the effects of tea gargling on influenza infection, and the clinical evidence is unclear. Also there have been no studies reported on the gargling effects with tea catechin extracts on the prevention of influenza infection.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* aged 20 to 65 years old
* obtained written informed concent before participation
* inoculated with influenza vaccine before entering the study

Exclusion Criteria:

* other gargling except water during the study
* possessing tea allergy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2005-11; Study Completion 2006-04

PRIMARY OUTCOMES:
Incidence rates of influenza infection during the study

SECONDARY OUTCOMES:
severity of symptoms including complications and hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Yamada, MD, PhD, Principal Investigator — University of Shizuoka
Locations (3):
- Japan (3):
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Shizuoka General Hospial, Shizuoka, Shizuoka
  - White Cross Nursing Home, Higashimurayama, Tokyo